CLINICAL TRIAL: NCT05497336
Title: An Open-label, Multicenter, Phase Ib/III Study of Efficacy and Safety of IBI351 in Combination With Cetuximab in Subjects With KRAS G12C Mutated Metastatic Colorectal Cancer
Brief Title: A Study of IBI351 in Combination With Cetuximab in Subjects With KRAS G12C Mutated Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI351B301
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI351+Cetuximab (Experimental): IBI351 recommended dose+Cetuximab 500mg/m2 IV Q2W
  Interventions: Drug: IBI351; Drug: Cetuximab
- IBI351 (Experimental): IBI351 recommended dose
  Interventions: Drug: IBI351

INTERVENTIONS:
Drug: IBI351 — IBI351 is administered orally
  Other Names: GFH925
Drug: Cetuximab — Cetuximab is administered intravenously
  Other Names: Erbitux
  Arms: IBI351+Cetuximab

SUMMARY:
Phase 1b consists of combined dose escalation phase and dose expansion phase. Phase 3 study will compare efficacy and safety of IBI351 combined with cetuximab versus chemotherapy in treatment of KRAS G12C-mutated metastatic colorectal cancer

DETAILED DESCRIPTION:
A Phase 1b study of the safety, tolerability and preliminary efficacy of IBI351 combined with cetuximab in the treatment of KRAS G12C mutant metastatic colorectal cancer will be conducted based on recommended dose of IBI351, which consists of combined dose escalation phase and dose expansion phase. After confirming the efficacy and safety of IBI351 combined with cetuximab in Phase Ib, an open-label Phase 3 study of the efficacy and safety of IBI351 combined with cetuximab versus oxaliplatin-based mFOLFOX6 regimen or irinotecan-based FOLFIRI with or without bevacizumab in treatment of KRAS G12C-mutated metastatic colorectal cancer will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. male or female subjects, ≥ 18 years and ≤ 75 years
2. have documentation of KRAS G12C mutation
3. at least one measurable lesion per RECISTv1.1
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
5. life expectancy of >12 weeks, in the opinion of the investigator

Exclusion Criteria:

1. history of deep venous thrombosis or any other serious thromboembolism within 3 months prior to enrollment..
2. history of radiation-induced pneumonitis, idiopathic pneumonia, active pneumonia, pulmonary fibrosis, diffuse pulmonary interstitial disease, or organizing pneumonia.
3. surgical procedures (excluding needle biopsy) performed within 28 days prior to enrollment that may affect the dosing or study assessments in this study.
4. received therapeutic or palliative radiation therapy within 14 days prior to enrollment
5. pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs (Dose-limiting Toxicity) in the Combined Dose Escalation Phase | 28 days during the first 4-week cycle
Objective response rate (ORR) | Up to 1 year

SECONDARY OUTCOMES:
incidence of serious treatment-emergent AEs (TEAEs) , treatment-related adverse event(TRAE), adverse events (SAEs) | up to 30 days after the last administration
Number of participants with abnormality in vital signs | up to 30 days after the last administration
Number of participants with abnormality in hematology parameters | up to 30 days after the last administration
Number of participants with abnormality in clinical chemistry parameters | up to 30 days after the last administration
Number of participants with abnormality in routine urinalysis parameters | up to 30 days after the last administration
Number of participants with abnormality in ECG parameters | up to 30 days after the last administration

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No